CLINICAL TRIAL: NCT02089542
Title: Development of a Clinical Protocol to Use Intra-operative Near Infra-red Fluorescent Imaging in Thyroid and Parathyroid Surgery
Brief Title: Intra-operative Infra-red Fluorescent Imaging in Thyroid and Parathyroid Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STH17176
Record Dates: First submitted 2014-03-13; First posted 2014-03-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Total Thyroidectomy; Bilateral Neck Exploration for Primary Hyperparathyroidism
Keywords: thyroidectomy; parathyroid surgery; parathyroid identification; methylene blue; near infrared fluorescence; intraoperative imaging
MeSH Terms: interventions — Methylene Blue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MB and fluorescent imaging (Experimental): Single arm study for the development of a protocol stipulating the optimum dose and time to peak near infra-red fluorescence from intraoperative injection of low dose Methylthioninium chloride
  Interventions: Other: MB and fluorescent imaging

INTERVENTIONS:
Other: MB and fluorescent imaging — Single arm study for the development of a protocol stipulating the optimum dose and time to peak near infra-red fluorescence from intraoperative injection of low dose Methylthioninium chloride
  Other Names: Methylthioninium chloride; Fluobeam 700 near infra-red imaging device

SUMMARY:
Reliable identification of parathyroid glands is critical to the success of thyroid and parathyroid surgery. In thyroid surgery, inadvertent injury to parathyroid glands may cause temporary or permanent hypoparathyroidism (low calcium levels needing long term treatment). In parathyroid surgery, early identification of normal and/or enlarged parathyroid glands helps in deciding on the extent of surgery and increases the chances of postoperative normal calcium levels.

Methylene Blue (Methylthioninium chloride, MB) is a dye that when given intravenously in high doses, is taken up differently by thyroid and parathyroid tissue. It is currently used during parathyroid surgery by some surgeons to help identify enlarged parathyroid glands by visual examination alone. Such visual examination is unhelpful in the identification of 'normal' parathyroid tissue. MB exhibits fluorescent properties in the near-infrared range (light just beyond the visible spectrum). This can be picked up by an appropriate imaging system. This has potential to identify and differentiate between 'normal' parathyroid, 'abnormal' parathyroid and thyroid tissue during surgery.

The investigators have established the feasibility of the intra-operative use of a near infra-red fluorescent imaging device called Fluobeam® and demonstrated the ability of this device to pick up near infra-red fluorescence from human tissue after administration of intravenous MB. Animal experiments have shown that doses as low as 0.1mg/kg of MB given intravenously enable fluorescent visualisation of thyroid and parathyroid glands.

This study will aim to optimise the dose and timing of administration of MB in human thyroid and parathyroid surgery and to develop a protocol which would then subsequently be assessed for effectiveness in a multi-centred randomized controlled setting.

DETAILED DESCRIPTION:
Around 13,000 thyroid and parathyroid operations are performed per year in England for both benign and malignant disease. Reliable identification of parathyroid glands is critical to the success of thyroid and parathyroid surgery. In thyroid surgery, inadvertent injury to parathyroid glands may cause temporary or permanent hypoparathyroidism (low calcium levels needing long term treatment); the latter is associated with significant long term problems. In parathyroid surgery, early identification of normal and/or enlarged parathyroid glands helps in deciding on the extent of surgery and increases the chances of postoperative normal calcium levels.

Methylene Blue (Methylthioninium chloride, MB) is a dye that when given intravenously in high doses, is taken up differently by thyroid and parathyroid tissue. It is currently used during parathyroid surgery by some surgeons to help identify enlarged parathyroid glands by visual examination alone. At these doses, there is a risk of adverse effects from administration of MB. Such visual examination is unhelpful in the identification of 'normal' parathyroid tissue. MB is not currently used in surgery for thyroid pathologies. MB exhibits fluorescent properties in the near-infrared range (light just beyond the visible spectrum). This can be picked up by an appropriate imaging system. This has potential to identify and differentiate between 'normal' parathyroid, 'abnormal' parathyroid and thyroid tissue during surgery.

The investigators have established the feasibility of the intra-operative use of a near infra-red fluorescent imaging device called Fluobeam® and demonstrated the ability of this device to pick up near infra-red fluorescence from human tissue after administration of intravenous MB. Animal experiments have shown that doses as low as 0.1mg/kg of MB given intravenously enable fluorescent visualisation of thyroid and parathyroid glands.

This study will aim to optimise the dose and timing of administration of MB in human thyroid and parathyroid surgery and to develop a protocol which would then subsequently be assessed for effectiveness in a multi-centred randomized controlled setting.

ELIGIBILITY:
Inclusion Criteria:

-All patients undergoing either a total thyroidectomy or bilateral neck exploration for PHPT in Sheffield Teaching Hospitals NHS Foundation Trust

Exclusion Criteria:

* Patients undergoing re-do procedures
* Patients unable to understand spoken and written English
* Patients unable to give adequate informed consent
* Patients with a history of intolerance or sensitivity to MB
* Patients with known G6PD deficiency
* Patients on serotonin reuptake inhibitors
* Patients undergoing surgery for thyroglossal cyst and
* Patients undergoing thoracic exploration; either alone or in combination with a neck exploration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-10; Primary Completion 2016-06 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Optimum dose of Methylene Blue | 20 minutes
  Determine optimum dose of Methylene Blue that will enable fluorescence to be detected from the soft tissue structures in the neck

SECONDARY OUTCOMES:
Time to peak fluorescence | 20 minutes
  Time to peak fluorescence at varying doses of Methylene Blue will be assessed during the observation period, which will be a maximum of twenty minutes.

OTHER OUTCOMES:
Postoperative calcium status | up to 12 weeks of surgery
Serious adverse event | up to 30 days after surgery
  This will include any one of the following:
  1. Death
  2. A life-threatening adverse event
  3. Inpatient hospitalisation or prolongation of existing hospitalisation
  4. A disability / incapacity
  5. A congenital anomaly in the offspring of a participant The reporting period for Serious Adverse Events will be from the time of induction of anaesthetic until 30 days after the day of surgery. Important medical events that may not result in death, be life-threatening, or require hospitalisation may be considered a serious adverse event when, based upon appropriate medical judgment, they may jeopardize the patient or participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. All adverse events will be assessed for seriousness, expectedness and causality.

CONTACTS AND LOCATIONS:
Overall Officials: Saba Balasubramanian, MS FRCS PhD, Principal Investigator — University of Sheffield
Locations (1):
- Department of General Surgery, Sheffield, South Yorkshire, United Kingdom